CLINICAL TRIAL: NCT01823744
Title: A New Strategy to Analyze Gene-Nutrient Interaction in Children and Adolescents
Brief Title: Harmonized Micronutrient Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12.07.NIHS
Record Dates: First submitted 2013-03-26; First posted 2013-04-04 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Genomic
Keywords: micronutrient; genomic; SAM/SAH ratio
MeSH Terms: interventions — Vitamins; Minerals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- micronutrient supplementation (Experimental): All the enrolled subjects will recieve orally, onca a day, during school days a chocolate bar including vitamins and minerals.
  The micronitrient supplementation will be consumed over 6 weeks, 5 days/week.
  Interventions: Dietary Supplement: micronutrient supplementation

INTERVENTIONS:
Dietary Supplement: micronutrient supplementation
  Other Names: Nestrovit: white chocolate bar with vitamins and minerals

SUMMARY:
The purpose of this trial is to better define how individuals with different genetic make-ups will require different interventions to improve their methylation potential and nutrient status.

DETAILED DESCRIPTION:
Despite the increasing incidence of overweight and obesity among children, nutritional deficiencies are still a concern.

A low intake of vitamins and minerals is associated with a reduction in the antioxidant capacity. Some vitamins are associated with chronic diseases including overweight and obesity.

S-adenosylmethionine (SAM) and S-adenosylhomocysteine (SAH) are the substrate and product of essential reactions; the SAM:SAH ratio has been associated with health and is an indicator of cellular DNA methylation potential.

Low level of this ratio may affect short and long term health. In this explorative knowledge building open interventional study, subject to be enrolled are children or adolescents 9 to 13 years of age per year (n=180 per year, over 2 years). The study consists of 6 weeks nutritional intervention followed by a 6 weeks follow up.

In this study, genomics, proteomics, lipidomics analysis will be performed, in addition to biochemistry, hematology and vitamins analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children or adolescents 9 to 13 years of age.
* Clinically stable.
* Normal weight, overweight and obese.

Exclusion Criteria:

* Disease diagnosis.
* At least one episode of axillary temperature >37°C over the prior 15 days.
* Three or more episodes of liquid or semi-liquid stools over the prior 24 hours.
* Supplementation with vitamins and/or minerals.
* On a supervised diet for reducing weight or any other type of diet restriction.
* Currently participating or having participated in another clinical study during the last 4 weeks prior to the beginning of this study.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
SAM/SAH ratio | baseline and after 6 weeks of product intake
  Change from baseline in the correlation between the SAM/SAH ratio in erythrocytes, dietary intakes and, polymorphisms in genes associated with micronutrients

SECONDARY OUTCOMES:
SNP arrays, proteomics, metabolomics, micronutrient levels | baseline, after 6 weeks of product intake and after 6 weeks of follow up
  Composite secondary outome: extensive "omic" analysis and correlation of the data over the 3 timepoints
SAM/SAH ratio | after 6 weeks product intake and after 6 weeks of follow up
  Change between 6 weeks after product intake and 6 weeks of follow up in the correlation between the SAM/SAH ratio in erythrocytes, dietary intakes and, polymorphisms in genes associated with micronutrients

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Pontes Monteiro, Profa. Dra., Principal Investigator — Campus Universitário USP, Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto
Locations (1):
- Campus Universitário USP, Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil